CLINICAL TRIAL: NCT02066454
Title: Evaluation of the Use of an Oral Direct Anti-Xa Anticoagulant, Apixaban, in Prevention of Venous Thromboembolic Disease in Patients Treated With IMiDs During Myeloma : a Pilot Study
Brief Title: Evaluation of the Use of Apixaban in Prevnetion of Thromboembolic Disease in Patients With Myeloma Trated With iMiDs
Acronym: MYELAXAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCIC 1320; 2013-003190-99 (EudraCT Number)
Record Dates: First submitted 2014-02-14; First posted 2014-02-19 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2015-03

CONDITIONS: Myeloma; Venous Thromboembolism
Keywords: myeloma; antiXa anticoagulant; venous thromboembolic disease; iMiDs
MeSH Terms: conditions — Neoplasms, Plasma Cell; Venous Thromboembolism | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apixaban (Experimental): oral direct anti-Xa anticoagulant
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — 2.5mg x 2 per day during 6 months
  Other Names: oral direct anti-Xa anticoagulant

SUMMARY:
To evaluate:

* the incidence of venous thromboembolic event (VTE)
* the incidence of hemorrhagic complications, In a population of patients with myeloma who are treated with IMiDs and require thromboprophylaxis for 6 months, using an oral anti-Xa anticoagulant, Apixaban, in a preventive scheme, 2.5 mg x2/day

DETAILED DESCRIPTION:
MYELAXAT trial is multicentre, open trial which aims to evaluate the incidence of venous thromboembolic event (VTE) and the incidence of hemorrhagic complications. All patients with Myeloma treated with iMiDs and require thromboprophylaxis for 6 months, using an oral anti-Xa anticoagulant, Apixaban, in a preventive scheme, 2.5 mg x2/day

ELIGIBILITY:
Inclusion Criteria:

* Patients (men/women) aged more than 18 years
* All consecutive patients, with myeloma, in first-line treatment or in relapse, who are treated - With IMiDs (MPT, Melphalan -Prednisone -Thalidomide ; Lenalidomide - Dexamethasone).

AND

- who require prevention of venous thromboembolic events with Aspirin or Low molecular Weight Heparin (LMWH) for a minimum duration of 6 months At least, 2/3 of patients will be treated with Lenalidomide-Dexamethasone.

* Written informed consent
* Patients affiliated to the French social security system or equivalent

Exclusion Criteria:

* Patient who needs curative anticoagulant treatment (heparin, LMWH, vitamin K antagonists, Dabigatran, Rivaroxaban, Apixaban) for an associated disorder (mechanical valve, atrial fibrillation or venous thromboembolic disease in the previous 6 months).
* Patient who needs preventive treatment with an anticoagulant in a post-operative context
* Patient who needs anti-platelet treatment (Aspirin, Clopidogrel, Prasugrel, Ticagrelor or dual anti-platelet therapy )
* Patient with active bleeding or at a high risk of bleeding (ulcer disease, intracranial bleeding in the previous 6 months, uncontrolled hypertension)
* Patient having undergone a surgical intervention within the past 30 days likely to expose them to an haemorrhagic risk
* Active hepatic disease (hepatitis, cirrhosis)
* Severe renal insufficiency (creatinine clearance using the Cockcroft equation < 30 ml/mn)
* Known allergic reaction to Apixaban
* Contraindication to the use of an anticoagulant treatment
* Prohibited concomitant treatment

  * inhibitors of CYP3A4 and P-gp : azole antimycotic agents (ketoconazole, itraconazole, voriconazole, posaconazole), inhibitors of HIV protease (ritonavir, indinavir, nelfinavir, atazanavir, saquinavir), specific macrolide antibiotics (clarithromycine, telithromycine)
  * other antithrombotic treatment : salicylate derivates (aspirin, products containing aspirin), antiplatelet therapy, heparin (unfractionated heparin, low molecular weight heparin, danaparoide sodique, fondaparinux), hirudines, oral anticoagulants (vitamin K antagonists, rivaroxaban, dabigatran)
* Patient with AST or ALT rate > 3 times upper limit of normal
* Patient with Bilirubin rate > 1.5 times upper limit of normal
* Patient with Platelets rate < 75 G/l
* Patient with Creatinine Clearance (Cockcroft) < 30 ml/mn
* Incidental finding of a proximal Deep Venous Thrombosis on the screening ultrasound
* Patients refusing or unable to give a written consent of information
* Patient unable to comply with the protocol requirement, in the investigator's opinion
* Life expectancy less than 6 months
* Incarcerated patients
* Pregnancy or possibility of pregnancy within 6 months
* Females of childbearing potential without reliable contraception
* Ecog > 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2016-07-12 (Actual); Study Completion 2016-07-12 (Actual)

PRIMARY OUTCOMES:
Total VTE and VTE-related death. Major and clinically relevant non major bleeding - Major and clinically relevant non major bleeding, defined according to International Society of Thrombosis and haemostasis | 7 months
  Total VTE (fatal or non fatal pulmonary embolism, symptomatic distal or proximal DVT of lower limbs, and asymptomatic proximal DVT detected by bilateral compression ultrasound) and VTE-related death.
  - Major and clinically relevant non major bleeding, defined according to International Society of Thrombosis and haemostasis

SECONDARY OUTCOMES:
incidence of venous thromboembolic complications | 7 months
  incidence of venous thromboembolic complications, symptomatic and asymptomatic, according to the thrombotic risk stratification of patients (low or high risk)
incidence of venous thromboembolic complications | 7 months
  incidence of venous thromboembolic complications, symptomatic and asymptomatic, according to the time of treatment with iMiDs (diagnosis or relapse)
incidence of major and clinically relevant non major bleeding | 7 months
  incidence of major and clinically relevant non major bleeding according to the thrombotic risk strtification of patients (low or high risk)
incidence of arterial cardiovascular events | 7 months
  incidence of arterial cardiovascular events (myocardial infarction, ischemic stroke, TIA)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte PEGOURIE, MD, Principal Investigator — Hospital University Grenoble; Gilles PERNOD, PHD, Principal Investigator — Hospital University Grenoble
Locations (19):
- France (19):
  - CHRA, Annecy
  - Ch La Cote Basque, Bayonne
  - Hia Percy, Clamart
  - Chu Hopital Henri Mondor, Créteil
  - Centre Hospitalier, Dunkirk
  - Chu Grenoble, Grenoble
  - Chd Vendee, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - Hopital St Vincent - Ghicl, Lille
  - Chru Hopital Huriez, Lille
  - Centre Leon Berard, Lyon
  - Groupe Hospitalier Du Havre, Montivilliers
  - Hopital de L'Archet, Nice
  - Hopital Pitie Salpetriere, Paris
  - Chu Bordeaux, Pessac
  - Ch de Perigueux, Périgueux
  - Ch Lyon Sud, Pierre-Bénite
  - Chu Poitiers, Poitiers
  - Chru de Tours, Tours

REFERENCES:
- [Background] Agnelli G, Buller HR, Cohen A, Curto M, Gallus AS, Johnson M, Porcari A, Raskob GE, Weitz JI; AMPLIFY-EXT Investigators. Apixaban for extended treatment of venous thromboembolism. N Engl J Med. 2013 Feb 21;368(8):699-708. doi: 10.1056/NEJMoa1207541. Epub 2012 Dec 8. PMID 23216615
- [Background] Anagnostopoulos A, Weber D, Rankin K, Delasalle K, Alexanian R. Thalidomide and dexamethasone for resistant multiple myeloma. Br J Haematol. 2003 Jun;121(5):768-71. doi: 10.1046/j.1365-2141.2003.04345.x. PMID 12780791
- [Background] Attal M, Lauwers-Cances V, Marit G, Caillot D, Moreau P, Facon T, Stoppa AM, Hulin C, Benboubker L, Garderet L, Decaux O, Leyvraz S, Vekemans MC, Voillat L, Michallet M, Pegourie B, Dumontet C, Roussel M, Leleu X, Mathiot C, Payen C, Avet-Loiseau H, Harousseau JL; IFM Investigators. Lenalidomide maintenance after stem-cell transplantation for multiple myeloma. N Engl J Med. 2012 May 10;366(19):1782-91. doi: 10.1056/NEJMoa1114138. PMID 22571202
- [Background] Barlogie B, Desikan R, Eddlemon P, Spencer T, Zeldis J, Munshi N, Badros A, Zangari M, Anaissie E, Epstein J, Shaughnessy J, Ayers D, Spoon D, Tricot G. Extended survival in advanced and refractory multiple myeloma after single-agent thalidomide: identification of prognostic factors in a phase 2 study of 169 patients. Blood. 2001 Jul 15;98(2):492-4. doi: 10.1182/blood.v98.2.492. PMID 11435324
- [Background] Baz R, Li L, Kottke-Marchant K, Srkalovic G, McGowan B, Yiannaki E, Karam MA, Faiman B, Jawde RA, Andresen S, Zeldis J, Hussein MA. The role of aspirin in the prevention of thrombotic complications of thalidomide and anthracycline-based chemotherapy for multiple myeloma. Mayo Clin Proc. 2005 Dec;80(12):1568-74. doi: 10.4065/80.12.1568. PMID 16342649
- [Background] Blom JW, Doggen CJ, Osanto S, Rosendaal FR. Malignancies, prothrombotic mutations, and the risk of venous thrombosis. JAMA. 2005 Feb 9;293(6):715-22. doi: 10.1001/jama.293.6.715. PMID 15701913
- [Background] Carrier M, Le Gal G, Tay J, Wu C, Lee AY. Rates of venous thromboembolism in multiple myeloma patients undergoing immunomodulatory therapy with thalidomide or lenalidomide: a systematic review and meta-analysis. J Thromb Haemost. 2011 Apr;9(4):653-63. doi: 10.1111/j.1538-7836.2011.04215.x. PMID 21255254
- [Background] Cavo M, Zamagni E, Tosi P, Cellini C, Cangini D, Tacchetti P, Testoni N, Tonelli M, de Vivo A, Palareti G, Tura S, Baccarani M. First-line therapy with thalidomide and dexamethasone in preparation for autologous stem cell transplantation for multiple myeloma. Haematologica. 2004 Jul;89(7):826-31. PMID 15257934
- [Background] Chen C, Reece DE, Siegel D, Niesvizky R, Boccia RV, Stadtmauer EA, Abonour R, Richardson P, Matous J, Kumar S, Bahlis NJ, Alsina M, Vescio R, Coutre SE, Pietronigro D, Knight RD, Zeldis JB, Rajkumar V. Expanded safety experience with lenalidomide plus dexamethasone in relapsed or refractory multiple myeloma. Br J Haematol. 2009 Jul;146(2):164-70. doi: 10.1111/j.1365-2141.2009.07728.x. Epub 2009 May 26. PMID 19545290
- [Background] Cohen AT, Davidson BL, Gallus AS, Lassen MR, Prins MH, Tomkowski W, Turpie AG, Egberts JF, Lensing AW; ARTEMIS Investigators. Efficacy and safety of fondaparinux for the prevention of venous thromboembolism in older acute medical patients: randomised placebo controlled trial. BMJ. 2006 Feb 11;332(7537):325-9. doi: 10.1136/bmj.38733.466748.7C. Epub 2006 Jan 26. PMID 16439370
- [Background] Cohen AT, Spiro TE, Buller HR, Haskell L, Hu D, Hull R, Mebazaa A, Merli G, Schellong S, Spyropoulos AC, Tapson V; MAGELLAN Investigators. Rivaroxaban for thromboprophylaxis in acutely ill medical patients. N Engl J Med. 2013 Feb 7;368(6):513-23. doi: 10.1056/NEJMoa1111096. PMID 23388003
- [Background] Connolly SJ, Eikelboom J, Joyner C, Diener HC, Hart R, Golitsyn S, Flaker G, Avezum A, Hohnloser SH, Diaz R, Talajic M, Zhu J, Pais P, Budaj A, Parkhomenko A, Jansky P, Commerford P, Tan RS, Sim KH, Lewis BS, Van Mieghem W, Lip GY, Kim JH, Lanas-Zanetti F, Gonzalez-Hermosillo A, Dans AL, Munawar M, O'Donnell M, Lawrence J, Lewis G, Afzal R, Yusuf S; AVERROES Steering Committee and Investigators. Apixaban in patients with atrial fibrillation. N Engl J Med. 2011 Mar 3;364(9):806-17. doi: 10.1056/NEJMoa1007432. Epub 2011 Feb 10. PMID 21309657
- [Background] Dimopoulos M, Spencer A, Attal M, Prince HM, Harousseau JL, Dmoszynska A, San Miguel J, Hellmann A, Facon T, Foa R, Corso A, Masliak Z, Olesnyckyj M, Yu Z, Patin J, Zeldis JB, Knight RD; Multiple Myeloma (010) Study Investigators. Lenalidomide plus dexamethasone for relapsed or refractory multiple myeloma. N Engl J Med. 2007 Nov 22;357(21):2123-32. doi: 10.1056/NEJMoa070594. PMID 18032762
- [Background] Facon T, Mary JY, Hulin C, Benboubker L, Attal M, Pegourie B, Renaud M, Harousseau JL, Guillerm G, Chaleteix C, Dib M, Voillat L, Maisonneuve H, Troncy J, Dorvaux V, Monconduit M, Martin C, Casassus P, Jaubert J, Jardel H, Doyen C, Kolb B, Anglaret B, Grosbois B, Yakoub-Agha I, Mathiot C, Avet-Loiseau H; Intergroupe Francophone du Myelome. Melphalan and prednisone plus thalidomide versus melphalan and prednisone alone or reduced-intensity autologous stem cell transplantation in elderly patients with multiple myeloma (IFM 99-06): a randomised trial. Lancet. 2007 Oct 6;370(9594):1209-18. doi: 10.1016/S0140-6736(07)61537-2. PMID 17920916
- [Background] Goldhaber SZ, Leizorovicz A, Kakkar AK, Haas SK, Merli G, Knabb RM, Weitz JI; ADOPT Trial Investigators. Apixaban versus enoxaparin for thromboprophylaxis in medically ill patients. N Engl J Med. 2011 Dec 8;365(23):2167-77. doi: 10.1056/NEJMoa1110899. Epub 2011 Nov 13. PMID 22077144
- [Background] Heit JA, Silverstein MD, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ 3rd. Risk factors for deep vein thrombosis and pulmonary embolism: a population-based case-control study. Arch Intern Med. 2000 Mar 27;160(6):809-15. doi: 10.1001/archinte.160.6.809. PMID 10737280
- [Background] Hussein MA. Thromboembolism risk reduction in multiple myeloma patients treated with immunomodulatory drug combinations. Thromb Haemost. 2006 Jun;95(6):924-30. doi: 10.1160/TH06-02-0080. PMID 16732369
- [Background] Johnson DC, Corthals S, Ramos C, Hoering A, Cocks K, Dickens NJ, Haessler J, Goldschmidt H, Child JA, Bell SE, Jackson G, Baris D, Rajkumar SV, Davies FE, Durie BG, Crowley J, Sonneveld P, Van Ness B, Morgan GJ. Genetic associations with thalidomide mediated venous thrombotic events in myeloma identified using targeted genotyping. Blood. 2008 Dec 15;112(13):4924-34. doi: 10.1182/blood-2008-02-140434. Epub 2008 Sep 19. PMID 18805967
- [Background] Kristinsson SY, Pfeiffer RM, Bjorkholm M, Goldin LR, Schulman S, Blimark C, Mellqvist UH, Wahlin A, Turesson I, Landgren O. Arterial and venous thrombosis in monoclonal gammopathy of undetermined significance and multiple myeloma: a population-based study. Blood. 2010 Jun 17;115(24):4991-8. doi: 10.1182/blood-2009-11-252072. Epub 2010 Mar 18. PMID 20299513
- [Background] Larocca A, Cavallo F, Bringhen S, Di Raimondo F, Falanga A, Evangelista A, Cavalli M, Stanevsky A, Corradini P, Pezzatti S, Patriarca F, Cavo M, Peccatori J, Catalano L, Carella AM, Cafro AM, Siniscalchi A, Crippa C, Petrucci MT, Yehuda DB, Beggiato E, Di Toritto TC, Boccadoro M, Nagler A, Palumbo A. Aspirin or enoxaparin thromboprophylaxis for patients with newly diagnosed multiple myeloma treated with lenalidomide. Blood. 2012 Jan 26;119(4):933-9; quiz 1093. doi: 10.1182/blood-2011-03-344333. Epub 2011 Aug 11. PMID 21835953
- [Background] Lassen MR, Raskob GE, Gallus A, Pineo G, Chen D, Hornick P; ADVANCE-2 investigators. Apixaban versus enoxaparin for thromboprophylaxis after knee replacement (ADVANCE-2): a randomised double-blind trial. Lancet. 2010 Mar 6;375(9717):807-15. doi: 10.1016/S0140-6736(09)62125-5. PMID 20206776
- [Background] Leizorovicz A, Cohen AT, Turpie AG, Olsson CG, Vaitkus PT, Goldhaber SZ; PREVENT Medical Thromboprophylaxis Study Group. Randomized, placebo-controlled trial of dalteparin for the prevention of venous thromboembolism in acutely ill medical patients. Circulation. 2004 Aug 17;110(7):874-9. doi: 10.1161/01.CIR.0000138928.83266.24. Epub 2004 Aug 2. PMID 15289368
- [Background] Leleu X, Daley L, Rodon P et al. MELISSE : Etude Multicentrique Prospective Observationelle pour definir les Facteurs de Risques de Thrombose dans le Myelome traite par les IMiDs. Congrès SFH, Paris, Mars 2011.
- [Background] Levine MN, Gu C, Liebman HA, Escalante CP, Solymoss S, Deitchman D, Ramirez L, Julian J. A randomized phase II trial of apixaban for the prevention of thromboembolism in patients with metastatic cancer. J Thromb Haemost. 2012 May;10(5):807-14. doi: 10.1111/j.1538-7836.2012.04693.x. PMID 22409262
- [Background] Libourel EJ, Sonneveld P, van der Holt B, de Maat MP, Leebeek FW. High incidence of arterial thrombosis in young patients treated for multiple myeloma: results of a prospective cohort study. Blood. 2010 Jul 8;116(1):22-6. doi: 10.1182/blood-2009-12-257519. Epub 2010 Mar 25. PMID 20339094
- [Background] Lyman GH, Khorana AA, Falanga A, Clarke-Pearson D, Flowers C, Jahanzeb M, Kakkar A, Kuderer NM, Levine MN, Liebman H, Mendelson D, Raskob G, Somerfield MR, Thodiyil P, Trent D, Francis CW; American Society of Clinical Oncology. American Society of Clinical Oncology guideline: recommendations for venous thromboembolism prophylaxis and treatment in patients with cancer. J Clin Oncol. 2007 Dec 1;25(34):5490-505. doi: 10.1200/JCO.2007.14.1283. Epub 2007 Oct 29. PMID 17968019
- [Background] Mileshkin L, Biagi JJ, Mitchell P, Underhill C, Grigg A, Bell R, McKendrick J, Briggs P, Seymour JF, Lillie K, Smith JG, Zeldis JB, Prince HM. Multicenter phase 2 trial of thalidomide in relapsed/refractory multiple myeloma: adverse prognostic impact of advanced age. Blood. 2003 Jul 1;102(1):69-77. doi: 10.1182/blood-2002-09-2846. Epub 2003 Mar 13. PMID 12637329
- [Background] Minnema MC, Breitkreutz I, Auwerda JJ, van der Holt B, Cremer FW, van Marion AM, Westveer PH, Sonneveld P, Goldschmidt H, Lokhorst HM. Prevention of venous thromboembolism with low molecular-weight heparin in patients with multiple myeloma treated with thalidomide and chemotherapy. Leukemia. 2004 Dec;18(12):2044-6. doi: 10.1038/sj.leu.2403533. No abstract available. PMID 15470485
- [Background] Neben K, Moehler T, Benner A, Kraemer A, Egerer G, Ho AD, Goldschmidt H. Dose-dependent effect of thalidomide on overall survival in relapsed multiple myeloma. Clin Cancer Res. 2002 Nov;8(11):3377-82. PMID 12429624
- [Background] Osman K, Comenzo R, Rajkumar SV. Deep venous thrombosis and thalidomide therapy for multiple myeloma. N Engl J Med. 2001 Jun 21;344(25):1951-2. doi: 10.1056/NEJM200106213442516. No abstract available. PMID 11419443
- [Background] Palumbo A, Bertola A, Falco P, Rosato R, Cavallo F, Giaccone L, Bringhen S, Musto P, Pregno P, Caravita T, Ciccone G, Boccadoro M. Efficacy of low-dose thalidomide and dexamethasone as first salvage regimen in multiple myeloma. Hematol J. 2004;5(4):318-24. doi: 10.1038/sj.thj.6200403. PMID 15297848
- [Background] Palumbo A, Bringhen S, Caravita T, Merla E, Capparella V, Callea V, Cangialosi C, Grasso M, Rossini F, Galli M, Catalano L, Zamagni E, Petrucci MT, De Stefano V, Ceccarelli M, Ambrosini MT, Avonto I, Falco P, Ciccone G, Liberati AM, Musto P, Boccadoro M; Italian Multiple Myeloma Network, GIMEMA. Oral melphalan and prednisone chemotherapy plus thalidomide compared with melphalan and prednisone alone in elderly patients with multiple myeloma: randomised controlled trial. Lancet. 2006 Mar 11;367(9513):825-31. doi: 10.1016/S0140-6736(06)68338-4. PMID 16530576
- [Background] Palumbo A, Rus C, Zeldis JB, Rodeghiero F, Boccadoro M; Italian Multiple Myeloma Network, Gimema. Enoxaparin or aspirin for the prevention of recurrent thromboembolism in newly diagnosed myeloma patients treated with melphalan and prednisone plus thalidomide or lenalidomide. J Thromb Haemost. 2006 Aug;4(8):1842-5. doi: 10.1111/j.1538-7836.2006.02059.x. No abstract available. PMID 16879233
- [Background] Palumbo A, Rajkumar SV, Dimopoulos MA, Richardson PG, San Miguel J, Barlogie B, Harousseau J, Zonder JA, Cavo M, Zangari M, Attal M, Belch A, Knop S, Joshua D, Sezer O, Ludwig H, Vesole D, Blade J, Kyle R, Westin J, Weber D, Bringhen S, Niesvizky R, Waage A, von Lilienfeld-Toal M, Lonial S, Morgan GJ, Orlowski RZ, Shimizu K, Anderson KC, Boccadoro M, Durie BG, Sonneveld P, Hussein MA; International Myeloma Working Group. Prevention of thalidomide- and lenalidomide-associated thrombosis in myeloma. Leukemia. 2008 Feb;22(2):414-23. doi: 10.1038/sj.leu.2405062. Epub 2007 Dec 20. PMID 18094721
- [Background] Palumbo A, Bringhen S, Liberati AM, Caravita T, Falcone A, Callea V, Montanaro M, Ria R, Capaldi A, Zambello R, Benevolo G, Derudas D, Dore F, Cavallo F, Gay F, Falco P, Ciccone G, Musto P, Cavo M, Boccadoro M. Oral melphalan, prednisone, and thalidomide in elderly patients with multiple myeloma: updated results of a randomized controlled trial. Blood. 2008 Oct 15;112(8):3107-14. doi: 10.1182/blood-2008-04-149427. Epub 2008 May 27. PMID 18505783
- [Background] Palumbo A, Davies F, Kropff M, Blade J, Delforge M, Leal da Costa F, Garcia Sanz R, Schey S, Facon T, Morgan G, Moreau P. Consensus guidelines for the optimal management of adverse events in newly diagnosed, transplant-ineligible patients receiving melphalan and prednisone in combination with thalidomide (MPT) for the treatment of multiple myeloma. Ann Hematol. 2010 Aug;89(8):803-11. doi: 10.1007/s00277-010-0925-1. Epub 2010 Mar 16. PMID 20232066
- [Background] Palumbo A, Cavo M, Bringhen S, Zamagni E, Romano A, Patriarca F, Rossi D, Gentilini F, Crippa C, Galli M, Nozzoli C, Ria R, Marasca R, Montefusco V, Baldini L, Elice F, Callea V, Pulini S, Carella AM, Zambello R, Benevolo G, Magarotto V, Tacchetti P, Pescosta N, Cellini C, Polloni C, Evangelista A, Caravita T, Morabito F, Offidani M, Tosi P, Boccadoro M. Aspirin, warfarin, or enoxaparin thromboprophylaxis in patients with multiple myeloma treated with thalidomide: a phase III, open-label, randomized trial. J Clin Oncol. 2011 Mar 10;29(8):986-93. doi: 10.1200/JCO.2010.31.6844. Epub 2011 Jan 31. PMID 21282540
- [Background] Pernod G, Albaladejo P, Godier A, Samama CM, Susen S, Gruel Y, Blais N, Fontana P, Cohen A, Llau JV, Rosencher N, Schved JF, de Maistre E, Samama MM, Mismetti P, Sie P; Working Group on Perioperative Haemostasis. Management of major bleeding complications and emergency surgery in patients on long-term treatment with direct oral anticoagulants, thrombin or factor-Xa inhibitors: proposals of the working group on perioperative haemostasis (GIHP) - March 2013. Arch Cardiovasc Dis. 2013 Jun-Jul;106(6-7):382-93. doi: 10.1016/j.acvd.2013.04.009. Epub 2013 Jun 25. PMID 23810130
- [Background] Rajkumar SV, Hayman S, Gertz MA, Dispenzieri A, Lacy MQ, Greipp PR, Geyer S, Iturria N, Fonseca R, Lust JA, Kyle RA, Witzig TE. Combination therapy with thalidomide plus dexamethasone for newly diagnosed myeloma. J Clin Oncol. 2002 Nov 1;20(21):4319-23. doi: 10.1200/JCO.2002.02.116. PMID 12409330
- [Background] Rajkumar SV, Gertz MA, Lacy MQ, Dispenzieri A, Fonseca R, Geyer SM, Iturria N, Kumar S, Lust JA, Kyle RA, Greipp PR, Witzig TE. Thalidomide as initial therapy for early-stage myeloma. Leukemia. 2003 Apr;17(4):775-9. doi: 10.1038/sj.leu.2402866. PMID 12682636
- [Background] Rajkumar SV, Hayman SR, Lacy MQ, Dispenzieri A, Geyer SM, Kabat B, Zeldenrust SR, Kumar S, Greipp PR, Fonseca R, Lust JA, Russell SJ, Kyle RA, Witzig TE, Gertz MA. Combination therapy with lenalidomide plus dexamethasone (Rev/Dex) for newly diagnosed myeloma. Blood. 2005 Dec 15;106(13):4050-3. doi: 10.1182/blood-2005-07-2817. Epub 2005 Aug 23. PMID 16118317
- [Background] Rajkumar SV, Blood E, Vesole D, Fonseca R, Greipp PR; Eastern Cooperative Oncology Group. Phase III clinical trial of thalidomide plus dexamethasone compared with dexamethasone alone in newly diagnosed multiple myeloma: a clinical trial coordinated by the Eastern Cooperative Oncology Group. J Clin Oncol. 2006 Jan 20;24(3):431-6. doi: 10.1200/JCO.2005.03.0221. Epub 2005 Dec 19. PMID 16365178
- [Background] Rajkumar SV, Jacobus S, Callander NS, Fonseca R, Vesole DH, Williams ME, Abonour R, Siegel DS, Katz M, Greipp PR; Eastern Cooperative Oncology Group. Lenalidomide plus high-dose dexamethasone versus lenalidomide plus low-dose dexamethasone as initial therapy for newly diagnosed multiple myeloma: an open-label randomised controlled trial. Lancet Oncol. 2010 Jan;11(1):29-37. doi: 10.1016/S1470-2045(09)70284-0. Epub 2009 Oct 21. PMID 19853510
- [Background] Samama MM, Cohen AT, Darmon JY, Desjardins L, Eldor A, Janbon C, Leizorovicz A, Nguyen H, Olsson CG, Turpie AG, Weisslinger N. A comparison of enoxaparin with placebo for the prevention of venous thromboembolism in acutely ill medical patients. Prophylaxis in Medical Patients with Enoxaparin Study Group. N Engl J Med. 1999 Sep 9;341(11):793-800. doi: 10.1056/NEJM199909093411103. PMID 10477777
- [Background] Samama CM. [Perioperative venous thromboembolism prophylaxis: short review and recommendations]. Ann Fr Anesth Reanim. 2008 Dec;27 Suppl 3:S2-8. doi: 10.1016/S0750-7658(08)75140-2. French. PMID 19185783
- [Background] Schey SA, Cavenagh J, Johnson R, Child JA, Oakervee H, Jones RW. An UK myeloma forum phase II study of thalidomide; long term follow-up and recommendations for treatment. Leuk Res. 2003 Oct;27(10):909-14. doi: 10.1016/s0145-2126(03)00027-4. PMID 12860011
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Schutt P, Ebeling P, Buttkereit U, Brandhorst D, Opalka B, Hoiczyk M, Flasshove M, Hense J, Bojko P, Metz K, Moritz T, Seeber S, Nowrousian MR. Thalidomide in combination with vincristine, epirubicin and dexamethasone (VED) for previously untreated patients with multiple myeloma. Eur J Haematol. 2005 Jan;74(1):40-6. doi: 10.1111/j.1600-0609.2004.00349.x. PMID 15613105
- [Background] Sidra G, Williams CD, Russell NH, Zaman S, Myers B, Byrne JL. Combination chemotherapy with cyclophosphamide, thalidomide and dexamethasone for patients with refractory, newly diagnosed or relapsed myeloma. Haematologica. 2006 Jun;91(6):862-3. PMID 16769594
- [Background] Sie P, Samama CM, Godier A, Rosencher N, Steib A, Llau JV, Van der Linden P, Pernod G, Lecompte T, Gouin-Thibault I, Albaladejo P; Working Group on Perioperative Haemostasis; French Study Group on Thrombosis and Haemostasis. Surgery and invasive procedures in patients on long-term treatment with direct oral anticoagulants: thrombin or factor-Xa inhibitors. Recommendations of the Working Group on Perioperative Haemostasis and the French Study Group on Thrombosis and Haemostasis. Arch Cardiovasc Dis. 2011 Dec;104(12):669-76. doi: 10.1016/j.acvd.2011.09.001. Epub 2011 Oct 29. PMID 22152517
- [Background] Singhal S, Mehta J, Desikan R, Ayers D, Roberson P, Eddlemon P, Munshi N, Anaissie E, Wilson C, Dhodapkar M, Zeddis J, Barlogie B. Antitumor activity of thalidomide in refractory multiple myeloma. N Engl J Med. 1999 Nov 18;341(21):1565-71. doi: 10.1056/NEJM199911183412102. PMID 10564685
- [Background] Sjalander A, Jansson JH, Bergqvist D, Eriksson H, Carlberg B, Svensson P. Efficacy and safety of anticoagulant prophylaxis to prevent venous thromboembolism in acutely ill medical inpatients: a meta-analysis. J Intern Med. 2008 Jan;263(1):52-60. doi: 10.1111/j.1365-2796.2007.01878.x. PMID 18088252
- [Background] Srkalovic G, Cameron MG, Rybicki L, Deitcher SR, Kattke-Marchant K, Hussein MA. Monoclonal gammopathy of undetermined significance and multiple myeloma are associated with an increased incidence of venothromboembolic disease. Cancer. 2004 Aug 1;101(3):558-66. doi: 10.1002/cncr.20405. PMID 15274069
- [Background] Turpie AG, Lassen MR, Eriksson BI, Gent M, Berkowitz SD, Misselwitz F, Bandel TJ, Homering M, Westermeier T, Kakkar AK. Rivaroxaban for the prevention of venous thromboembolism after hip or knee arthroplasty. Pooled analysis of four studies. Thromb Haemost. 2011 Mar;105(3):444-53. doi: 10.1160/TH10-09-0601. Epub 2010 Dec 6. PMID 21136019
- [Background] Weber D, Rankin K, Gavino M, Delasalle K, Alexanian R. Thalidomide alone or with dexamethasone for previously untreated multiple myeloma. J Clin Oncol. 2003 Jan 1;21(1):16-9. doi: 10.1200/JCO.2003.03.139. PMID 12506164
- [Background] Wu P, Davies FE, Horton C, Jenner MW, Krishnan B, Alvares CL, Saso R, McCormack R, Dines S, Treleaven JG, Potter MN, Ethell ME, Morgan GJ. The combination of cyclophosphomide, thalidomide and dexamethasone is an effective alternative to cyclophosphamide - vincristine - doxorubicin - methylprednisolone as induction chemotherapy prior to autologous transplantation for multiple myeloma: a case-matched analysis. Leuk Lymphoma. 2006 Nov;47(11):2335-8. doi: 10.1080/10428190600821955. PMID 17107906
- [Background] Zangari M, Anaissie E, Barlogie B, Badros A, Desikan R, Gopal AV, Morris C, Toor A, Siegel E, Fink L, Tricot G. Increased risk of deep-vein thrombosis in patients with multiple myeloma receiving thalidomide and chemotherapy. Blood. 2001 Sep 1;98(5):1614-5. doi: 10.1182/blood.v98.5.1614. PMID 11520815
- [Background] Zangari M, Siegel E, Barlogie B, Anaissie E, Saghafifar F, Fassas A, Morris C, Fink L, Tricot G. Thrombogenic activity of doxorubicin in myeloma patients receiving thalidomide: implications for therapy. Blood. 2002 Aug 15;100(4):1168-71. doi: 10.1182/blood-2002-01-0335. PMID 12149193
- [Background] Zangari M, Barlogie B, Anaissie E, Saghafifar F, Eddlemon P, Jacobson J, Lee CK, Thertulien R, Talamo G, Thomas T, Van Rhee F, Fassas A, Fink L, Tricot G. Deep vein thrombosis in patients with multiple myeloma treated with thalidomide and chemotherapy: effects of prophylactic and therapeutic anticoagulation. Br J Haematol. 2004 Sep;126(5):715-21. doi: 10.1111/j.1365-2141.2004.05078.x. PMID 15327525
- [Background] Zervas K, Dimopoulos MA, Hatzicharissi E, Anagnostopoulos A, Papaioannou M, Mitsouli Ch, Panagiotidis P, Korantzis J, Tzilianos M, Maniatis A; Greek Myeloma Study Group. Primary treatment of multiple myeloma with thalidomide, vincristine, liposomal doxorubicin and dexamethasone (T-VAD doxil): a phase II multicenter study. Ann Oncol. 2004 Jan;15(1):134-8. doi: 10.1093/annonc/mdh026. PMID 14679133
- [Background] Zonder JA, Barlogie B, Durie BG, McCoy J, Crowley J, Hussein MA. Thrombotic complications in patients with newly diagnosed multiple myeloma treated with lenalidomide and dexamethasone: benefit of aspirin prophylaxis. Blood. 2006 Jul 1;108(1):403; author reply 404. doi: 10.1182/blood-2006-01-0154. No abstract available. PMID 16790586
- [Background] Zonder JA, Crowley J, Hussein MA, Bolejack V, Moore DF Sr, Whittenberger BF, Abidi MH, Durie BG, Barlogie B. Lenalidomide and high-dose dexamethasone compared with dexamethasone as initial therapy for multiple myeloma: a randomized Southwest Oncology Group trial (S0232). Blood. 2010 Dec 23;116(26):5838-41. doi: 10.1182/blood-2010-08-303487. Epub 2010 Sep 27. PMID 20876454
- [Background] Zufferey P, Laporte S, Quenet S, Molliex S, Auboyer C, Decousus H, Mismetti P. Optimal low-molecular-weight heparin regimen in major orthopaedic surgery. A meta-analysis of randomised trials. Thromb Haemost. 2003 Oct;90(4):654-61. doi: 10.1160/TH03-02-0086. PMID 14515186
- [Result] Pegourie B, Karlin L, Benboubker L, Orsini-Piocelle F, Tiab M, Auger-Quittet S, Rodon P, Royer B, Leleu X, Bareau B, Cliquennois M, Fuzibet JG, Voog E, Belhadj-Merzoug K, Decaux O, Rey P, Slama B, Leyronnas C, Zarnitsky C, Boyle E, Bosson JL, Pernod G; IFM Group. Apixaban for the prevention of thromboembolism in immunomodulatory-treated myeloma patients: Myelaxat, a phase 2 pilot study. Am J Hematol. 2019 Jun;94(6):635-640. doi: 10.1002/ajh.25459. Epub 2019 Apr 1. PMID 30859608